CLINICAL TRIAL: NCT03161665
Title: A Pilot Study of Patient and Caregiver Participation Through an Educational Health Information Technology System ("BMT Roadmap") in the Context of Hematopoietic Cell Transplantation (Adult Protocol)
Brief Title: Patient and Caregiver Participation Through an Educational Health Information Technology System ("BMT Roadmap") in the Context of Hematopoietic Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2015.140; HUM00107014 (Other: University of Michigan)
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Patients Undergoing Bone Marrow Transplant (BMT)

STUDY DESIGN:
Intervention Model Description: The BMT Roadmap information system will be tested in 20 caregivers of patients undergoing autologous or allogeneic BMT and 20 patients undergoing autologous or allogeneic BMT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMT Roadmap (Experimental): The BMT Roadmap information system will be tested in 20 caregivers of patients undergoing autologous or allogeneic BMT and in 20 patients undergoing autologous or allogeneic BMT.
  Interventions: Other: BMT Roadmap

INTERVENTIONS:
Other: BMT Roadmap — The BMT Roadmap is a health IT System that has been developed for use on the Apple iPad® to give the patient and caregivers easy access to test results, current treatment and contact information to hopefully increase active participation and engagement in transplant care.

SUMMARY:
Hematopoietic cell transplantation (BMT), or commonly referred to as blood and marrow transplantation (BMT), is a potentially life-saving therapy for many malignant and non-malignant conditions. Despite advances over the past decade, which have led to improved outcomes, BMT remains an intense treatment modality often requiring prolonged inpatient--based care. While many patients endure the acute complications of the procedure, it is common for BMT patients and their caregivers to experience increased risk of financial and emotional burden, hospital readmission, and health service utilization. This highlights the importance of active involvement of BMT patients in their own health care (self--efficacy).

Given the intense nature of BMT, however, caregivers also play a critical role in the process and are a necessary component of proceeding with transplant. As such, caregiver activation on behalf of the patient plays a critical role in effective patient--caregiver-provider partnerships, which is increasingly recognized as the optimal model for health care delivery, particularly for those facing life--altering medical treatments. It is essential to develop effective strategies to enhance this partnership. Health information technology (IT)-mediated tools offer the potential to overcome constraints in health care delivery limited by provider time, complicated health information, and financial pressures. Significant gaps in knowledge exist on the use of health IT tools using low- cost and well- accepted delivery platforms in routine inpatient care, especially for high- risk or critically ill populations. We hypothesize that a tablet--based tool displaying personal health information could provide a platform to promote caregiver activation and enhance health communication.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited by BMT RN Coordinators and physicians prior to patient admission to the BMT Unit. Caregiver (age 18 years or older) of any patient eligible to undergo autologous or allogeneic BMT and any patient (age 18 years or older) eligible to undergo autologous or allogeneic BMT will be recruited during the "Pre-Transplant Work-up" stage in the outpatient setting.
* CAREGIVER PARTICIPANTS: Caregiver (age 18 years or older) of a patient who will be hospitalized to undergo first-time autologous (self) or allogeneic (alternative donor) BMT in the University of Michigan Mott Children's Hospital BMT Unit
* PATIENT PARTICIPANTS: Patients (age 18 years or older) who will be hospitalized to undergo first-time autologous or allogeneic BMT will be given the opportunity to assent/consent and participate in the study. With his/her permission, the patient will also be provided with their own iPad® BMT Roadmap information system to use. Qualitative interviews will be conducted in patients with their assent/consent.
* Ability to speak and read proficiently in English (the study's instruments have not been translated and validated in languages other than English)
* Willing and able to provide informed consent
* Willing to comply with study procedures and reporting requirements

Exclusion Criteria:

* Not willing and able to provide informed consent
* Not willing to comply with study procedures and reporting requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Caregivers Accrued | 5 months
  Feasibility of the study will be determined by demonstrating that accruing at least 20% of caregivers from the BMT patient population is possible.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Choi, M.D., M.S., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Fauer AJ, Hoodin F, Lalonde L, Errickson J, Runaas L, Churay T, Seyedsalehi S, Warfield C, Chappell G, Brookshire K, Chaar D, Shin JY, Byrd M, Magenau J, Hanauer DA, Choi SW. Impact of a health information technology tool addressing information needs of caregivers of adult and pediatric hematopoietic stem cell transplantation patients. Support Care Cancer. 2019 Jun;27(6):2103-2112. doi: 10.1007/s00520-018-4450-4. Epub 2018 Sep 20. PMID 30232587